CLINICAL TRIAL: NCT04508231
Title: Metabolic Consequences of Cross-sex Hormonal Treatment in Transgender Persons
Brief Title: Metabolic Consequences of Cross-sex Hormonal Treatment
Acronym: DysGeMet
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PI157
Record Dates: First submitted 2020-08-03; First posted 2020-08-11 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-07

CONDITIONS: Gender Dysphoria
MeSH Terms: conditions — Gender Dysphoria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hormonal treatment: The University Hospital in Nancy is an academic regional transgender referral center in Lorraine (France) and keeps a register of subjects available from 2004. The register at the time of the present study (February 2020) included 320 subjects who met diagnostic criteria for gender dysphoria and were seen regularly in the out-patient clinic at our department of endocrinology. Our investigation is a part of the regular care of subjects with gender dysphoria.
  Interventions: Other: Gender-affirming hormone therapy
- Controls: Data for control subjects are retrieved from medical records of healthy non-obese females and males who underwent an initial assessment for gender dysphoria in our department, but not yet receiving hormonal treatment at the time of the present study.

INTERVENTIONS:
Other: Gender-affirming hormone therapy — Gender-affirming hormone therapy according to the recommendations of the Endocrine Society
  Groups: Hormonal treatment

SUMMARY:
Retrospective study in a single academic regional transgender referral center. Analyse VAT, body composition and metabolic parameters in non-obese transgender subjects one year after starting gender-affirming hormone therapy and in controls

ELIGIBILITY:
Inclusion Criteria (retrospective analysis of available data as a part of the regular care of subjects with gender dysphoria. All measurements were made at the time of the routine follow-up visits)

* age >= 16 years (Tanner stage IV) and <= 50 years at the initiation of gender-affirming hormone therapy;
* BMI < 28 kg/m2 at the initiation of cross-sex hormonal treatment.

Exclusion Criteria:

* hormonal contraception
* previous gender-affirming hormonal treatment
* previous gender-affirming surgery
* recognized syndrome or chromosomal defect, known metabolic or inflammatory disease, skeletal dysplasia, or chronic corticosteroid treatment.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — Subjects who met diagnostic criteria for gender dysphoria (International Classification of Diseases 11th Revision. https://icdwhoint. 2018) and were seen regularly in the out-patient clinic at our department of endocrinology
Study Population: Subjects who met diagnostic criteria for gender dysphoria (International Classification of Diseases 11th Revision. https://icdwhoint. 2018) and were seen regularly in the out-patient clinic at our department of endocrinology
Sampling Method: Probability Sample
Enrollment: 98 (Estimated)
Dates: Start 2020-07-24 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Retrospective analysis of existing data collected as a part of the regular follow-up | Retrospective analysis of data between 2004 and 2019
  Retrospective analysis of existing data :Anthropometric parameters, including systolic blood pressure (SBP), diastolic blood pressure (DBP), body weight and height at fasting state, were measured in all subjects at the occasion of the routine follow-up visits. Body mass index (BMI) was calculated as body weight in kilograms divided by the height in meter squared (kg/m2). Body composition parameters, including lean mass (LM), total body fat (BF), android and gynoid fat, and bone mineral content, were determined using dual-energy X-Ray absorbtiometry (DXA) (GE-Healthcare Lunar iDXA system), biochemical and routine hormonal analysis

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Nancy, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Larose C, Samhani C, Consolandi P, Feigerlova E. Increase in visceral adipose tissue and altered metabolic profile in transgender men but not in transgender women one year after starting gender-affirming hormonal therapy. Endocrine. 2025 Sep;89(3):901-909. doi: 10.1007/s12020-025-04310-y. Epub 2025 Jun 10. PMID 40495044